CLINICAL TRIAL: NCT04671680
Title: Comparison of Continuous Non-Invasive Arterial Blood Pressure to Invasive Arterial Blood Pressure Measurement in Pregnant Women With Placenta Accreta
Brief Title: CNAP vs IABP in Pregnant Women With Placenta Accreta
Status: Terminated | Type: Observational
Why Stopped: Unable to obtain data from device
Sponsor: Beth Israel Deaconess Medical Center (Other)
Responsible Party: Principal Investigator, Phillip Hess, Associate Professor of Anaesthesia, Beth Israel Deaconess Medical Center
Other Study IDs: 2020P001099
Record Dates: First submitted 2020-11-30; First posted 2020-12-17 (Actual); Last update posted 2025-10-21 (Actual); Status verified 2025-10

CONDITIONS: Placenta Accreta; Blood Pressure; Hemorrhage; Hemorrhage, Postpartum
Keywords: Placenta Accreta; Non-Invasive Arterial Blood Pressure; Invasive Arterial Blood Pressure; Hemorrhage; Hemorrhage, Postpartum
MeSH Terms: conditions — Placenta Accreta; Hemorrhage; Postpartum Hemorrhage

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (1):
- Pregnant women with suspected placenta accreta: Pregnant women undergoing cesarean delivery with suspected placenta accreta spectrum.
  Interventions: Device: LiDCO CNAP Monitoring Equipment

INTERVENTIONS:
Device: LiDCO CNAP Monitoring Equipment — A continuous non-invasive arterial blood pressure monitor for rapidly changing hemodynamics.

SUMMARY:
The objective of this study is to investigate a technique to monitor blood pressure in women undergoing cesarean delivery with suspected placenta accreta spectrum. To achieve this objective, the investigators plan to conduct a prospective, observational study with the following aims:

Specific Aim 1: Compare concordance between the systolic (SBP), diastolic (DBP), and mean arterial blood pressure (MAP) readings from the continuous non-invasive arterial blood pressure (CNAP) and IABP at several discrete points throughout the procedure

Specific Aim 2: Determine the feasibility of using CNAP to aid in decision making by examining the parameters of volume responsiveness and arterial elastance at several discrete points throughout the procedure.

The investigators hypothesize that the investigators can obtain similar blood pressure monitoring using CNAP as compared to the gold standard IABP in women undergoing cesarean delivery with suspected placenta accreta.

DETAILED DESCRIPTION:
Study Overview This is a prospective, observational study.

Study Procedures Patients who meet inclusion criteria with no exclusions will be approached to provide written informed consent.

Enrolled patients will undergo the standard pre-operative evaluation and preparation for cesarean section with possible hysterectomy including evaluation by nursing, obstetrics and anesthesiology team, placement of 2 large bore IVs, arterial line placement and laboratory tests.

The patient will then be transported to the OR. In the OR the CNAP device will be placed on the patient's finger and be given a brief calibration period of 45 seconds. As per usual for this procedure, each patient will undergo combined spinal epidural anesthesia with our standard cesarean induction dose of hyperbaric intrathecal 0.75% bupivacaine 1.5ml, intrathecal fentanyl 25 micrograms and intrathecal morphine 250 micrograms. The patient will be moved to the supine position with left lateral uterine displacement. When a T6 sensory level to pinprick is achieved, surgery will be allowed to proceed. Throughout the surgery, the CNAP and IABP will take continuous reading of blood pressure and hemodynamic variable. Labs and additional fluid or blood may be given to the patient as clinically indicated, as is common for this procedure. Blood work will be obtained from the arterial line used for IABP, as is standard practice when an AIBP is in place. Other than the addition of the CNAP cuff, all other care will be per standard protocol for this procedure.

Data Collection In order to assess our primary and secondary outcomes, the investigators will be collecting CNAP and AIBP. Additional baseline characteristics including, but not limited to age, race, gender, BMI and comorbidities will be abstracted from the medical record. REDCap will be utilized for data collection and storage.

Primary Outcomes SBP, MAP, DBP reading from the CNAP and AIBP at several discrete points throughout the procedure.

Secondary Outcomes Additional comparisons of SBP, MAP, DBP measurements using CNAP to AIBP and NIBP, review of extrapolated data outputs including Stroke Volume, Systemic Vascular Resistance, Cardiac Output and Stroke Volume Variation from CNAP compared pulse pressure index from pulse oximetry and AIBP and their responsiveness to fluid bolus, subgroup analysis of CNAP and AIBP during times significant intravascular volume depletion (blood loss) or systemic vascular resistance change (after spinal anesthesia). Relevant clinical data will also be collected, including; demographic data, total estimated blood lose, total quantitative blood loss, length of hospital stay, routine lab results including; Hematocrit, Fibrinogen, coagulation tests, lactic acid, pH, base excess.

ELIGIBILITY:
Inclusion Criteria:

* Women aged 18-40 years old with pregnancy complicated by accreta spectrum undergoing elective, scheduled cesarean delivery and possible hysterectomy

Exclusion Criteria:

* Women aged <18
* Patients with cardiac arrhythmia
* Vascular pathologies of the upper limbs (recent vascular surgery, Reynaud's disease, vascular stenosis)
* Contraindication to neuraxial anesthesia
* Emergent cases
* Droplet or airborne precautions (as determined by BIDMC infection control policy)

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — This study will only enroll female patients given its focus on pregnancy-related complications
Study Population: Pregnant women undergoing cesarean delivery with suspected placenta accreta spectrum.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2021-01-15 (Actual); Primary Completion 2025-06-01 (Actual); Study Completion 2025-06-01 (Actual)

PRIMARY OUTCOMES:
Comparing concordance between MAP from the CNAP and AIBP | MAP will be measured continuously throughout the operative case, with an average case timeframe of 4-6 hours.
  Comparing concordance of systolic blood pressure, mean arterial blood pressure, and diastolic blood pressure readings captured from the continuous non-invasive arterial blood pressure measurements and invasive arterial blood pressure measurements.

SECONDARY OUTCOMES:
Additional Comparisons of SBP and DBP | SBP and DBP will be measured continuously throughout the operative case, with an average case timeframe of 4-6 hours.
Stroke Volume | Measured throughout the operative case, with an average case timeframe of 4-6 hours.
  Review of extrapolated data outputs to assess the volume of blood ejected from each ventricle due to the contraction of the heart muscle which compresses these ventricles, measurements in millilitres.
Systemic Vascular Resistance | Measured throughout the operative case, with an average case timeframe of 4-6 hours.
  Review of extrapolated data outputs to assess changes in the arterioles.
Cardiac Output | Measured throughout the operative case, with an average case timeframe of 4-6 hours.
  Review of extrapolated data outputs to assess heart rate product.
Stroke Volume Variation | Measured throughout the operative case, with an average case timeframe of 4-6 hours.
  Review of extrapolated data outputs assessing the change in the amount of blood ejected from the left ventricle into the aorta with each heartbeat
Subgroup analysis of CNAP and AIBP | Measured throughout the operative case, with an average case timeframe of 4-6 hours.
  Analysis of continuous non-invasive arterial blood pressure measurements and invasive arterial blood pressure measurements during times significant intravascular volume depletion (blood loss) or systemic vascular resistance change (after spinal anesthesia). This will include the above derived variables (SV, SVR, CO, SVV) and compare them to pulse pressure variation to assess potential value of these measures in the assessment volume depletion and fluid responsiveness.

CONTACTS AND LOCATIONS:
Overall Officials: John J. Kowalczyk, MD, Principal Investigator — Beth Israel Deaconess Medical Center
Locations (1):
- Beth Israel Deaconess Medical Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hamilton BE, Martin JA, Osterman MJ, Curtin SC, Matthews TJ. Births: Final Data for 2014. Natl Vital Stat Rep. 2015 Dec;64(12):1-64. PMID 26727629
- [Background] Creanga AA, Berg CJ, Syverson C, Seed K, Bruce FC, Callaghan WM. Pregnancy-related mortality in the United States, 2006-2010. Obstet Gynecol. 2015 Jan;125(1):5-12. doi: 10.1097/AOG.0000000000000564. PMID 25560097
- [Background] Creanga AA, Berg CJ, Ko JY, Farr SL, Tong VT, Bruce FC, Callaghan WM. Maternal mortality and morbidity in the United States: where are we now? J Womens Health (Larchmt). 2014 Jan;23(1):3-9. doi: 10.1089/jwh.2013.4617. PMID 24383493
- [Background] Chung E, Chen G, Alexander B, Cannesson M. Non-invasive continuous blood pressure monitoring: a review of current applications. Front Med. 2013 Mar;7(1):91-101. doi: 10.1007/s11684-013-0239-5. Epub 2013 Jan 23. PMID 23345112
- [Background] Stenglova A, Benes J. Continuous Non-Invasive Arterial Pressure Assessment during Surgery to Improve Outcome. Front Med (Lausanne). 2017 Nov 17;4:202. doi: 10.3389/fmed.2017.00202. eCollection 2017. PMID 29204425
- [Background] Maheshwari K, Khanna S, Bajracharya GR, Makarova N, Riter Q, Raza S, Cywinski JB, Argalious M, Kurz A, Sessler DI. A Randomized Trial of Continuous Noninvasive Blood Pressure Monitoring During Noncardiac Surgery. Anesth Analg. 2018 Aug;127(2):424-431. doi: 10.1213/ANE.0000000000003482. PMID 29916861
- [Background] Bartels K, Esper SA, Thiele RH. Blood Pressure Monitoring for the Anesthesiologist: A Practical Review. Anesth Analg. 2016 Jun;122(6):1866-79. doi: 10.1213/ANE.0000000000001340. PMID 27195632
- [Background] Rogge DE, Nicklas JY, Schon G, Grothe O, Haas SA, Reuter DA, Saugel B. Continuous Noninvasive Arterial Pressure Monitoring in Obese Patients During Bariatric Surgery: An Evaluation of the Vascular Unloading Technique (Clearsight system). Anesth Analg. 2019 Mar;128(3):477-483. doi: 10.1213/ANE.0000000000003943. PMID 30649073
- [Background] Sumiyoshi M, Maeda T, Miyazaki E, Hotta N, Sato H, Hamaguchi E, Kanazawa H, Ohnishi Y, Kamei M. Accuracy of the ClearSight system in patients undergoing abdominal aortic aneurysm surgery. J Anesth. 2019 Jun;33(3):364-371. doi: 10.1007/s00540-019-02632-6. Epub 2019 Mar 23. PMID 30904953
- [Background] Meidert AS, Nold JS, Hornung R, Paulus AC, Zwissler B, Czerner S. The impact of continuous non-invasive arterial blood pressure monitoring on blood pressure stability during general anaesthesia in orthopaedic patients: A randomised trial. Eur J Anaesthesiol. 2017 Nov;34(11):716-722. doi: 10.1097/EJA.0000000000000690. PMID 28922340
- [Background] Cecconi M, Monge Garcia MI, Gracia Romero M, Mellinghoff J, Caliandro F, Grounds RM, Rhodes A. The use of pulse pressure variation and stroke volume variation in spontaneously breathing patients to assess dynamic arterial elastance and to predict arterial pressure response to fluid administration. Anesth Analg. 2015 Jan;120(1):76-84. doi: 10.1213/ANE.0000000000000442. PMID 25230102
- [Background] Hohn A, Defosse JM, Becker S, Steffen C, Wappler F, Sakka SG. Non-invasive continuous arterial pressure monitoring with Nexfin does not sufficiently replace invasive measurements in critically ill patients. Br J Anaesth. 2013 Aug;111(2):178-84. doi: 10.1093/bja/aet023. Epub 2013 Mar 13. PMID 23485882
- [Background] Gupta D, Soskin V, Marjanovic M, Amhaz H, Mazumdar A. CONTINUOUS NON-INVASIVE ARTERIAL PRESSURE DEVICE AS AN ADJUNCT TO RECOGNIZE FLUCTUATING BLOOD PRESSURES DURING ELECTIVE CESAREAN SECTION UNDER SUBARACHNOID BLOCKADE (SAB). Middle East J Anaesthesiol. 2016 Feb;23(4):385-400. PMID 27382807